CLINICAL TRIAL: NCT02206815
Title: Safety of Ticagrelor Plus Warfarin Versus Clopidogrel+Aspirin+Warfarin in Patients With Persistent or Permanent Atrial Fibrillation and Undergoing PCI-S: A Randomized, Open, Controlled, Parallel Group, Multi-center Trial
Brief Title: Safety of "Ticagrelor+ Warfarin"in Comparison With "Clopidogrel+Aspirin+Warfarin"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genshan Ma (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Sponsor-Investigator, Genshan Ma, Genshan Ma, MD, PhD, Director of Cardiovascular Institute, Southeast University, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0256
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor+Warfarin (Active Comparator): Ticagrelor:Plain, round, yellow, film-coated tablet, 90mg; Warfarin:Plain, round, white, film-coated tablet, 2.5mg
  Interventions: Drug: Ticagrelor+Warfarin
- Clopidogrel+Aspirin+Warfarin (Active Comparator): Clopidogrel:Light red bisulfate tablets, containing one 75mg; Aspirin:Plain, round, white, film-coated tablet, 100mg; Warfarin:Plain, round, white, film-coated tablet, 2.5mg
  Interventions: Drug: Clopidogrel+Aspirin+Warfarin

INTERVENTIONS:
Drug: Ticagrelor+Warfarin — Ticagrelor 90mg/bid + Warfarin (maintain INR 2.0-2.5)
  Other Names: Double antithrombotic therapy
  Arms: Ticagrelor+Warfarin
Drug: Clopidogrel+Aspirin+Warfarin — Clopidogrel 75mg/day + Aspirin 100mg/day + Warfarin(maintain INR 2.0-2.5)
  Other Names: Triple antithrombotic therapy
  Arms: Clopidogrel+Aspirin+Warfarin

SUMMARY:
The aim of this study was to assess safety of antithrombotic drug ticagrelor plus oral anticoagulation adopted in persistent or permanent AF(Atrial fibrillation) patients（CHA2DS2VASc≥2） after PCI-S with specially regard to the occurrence of major bleeding complications. We hypothesized that baseline characteristics (ie age, anemia, previous major bleeding) and type of antithrombotic regimen could influence any bleeding events and the time of bleeding occurrence. We will test this hypothesis by comparing those AF patients who subsequently received double antithrombotic therapy (Ticagrelor + Warfarin) vs. triple antithrombotic therapy (Clopidogrel + Aspirin + Warfarin) after undergoing PCI-S.

DETAILED DESCRIPTION:
Currently, the optimal antithrombotic treatment of AF patients with indication for long-term oral anticoagulation undergoing PCI-S is unknown. The randomized trials to assess the best antithrombotic regimen in this setting and the management of this population are challenging. It poses imperative demands for future prospective randomized studies to define the optimal antithrombotic regimen in patients requiring chronic anticoagulation undergoing coronary stenting. Additionally, the vast majority of current clinical studies about antithrombotic therapy for atrial fibrillation together with PCI were retrospectively analysis to date ,whereas the prospective studies are rare and urgently needed

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in this study and signed an informed consent form;
* Men or non-pregnant women ≥ 18 and ≤75 years of age;
* Lesion is located in a coronary artery and the need for coronary drug-eluting stent implantation;
* Patients with persistent or permanent atrial fibrillation;
* Score of CHA2DS2VASc≥2.

Exclusion Criteria:

* Severe liver and kidney diseases (GFR<60 ml/min/1.73m2 or CTP≥6 score);
* Moderate to severe hypertension (after standard antihypertensive therapy, blood pressure higher than 160/100mmHg);
* Patients with hemodynamic or electrical instability (including shock);
* Coagulation disorders associated with significant bleeding tendency (eg, hypersensitivity, active bleeding, moderate or severe liver disease, history of previous intracranial bleed, GI bleed within the past 6 months, major surgery within 30 days);
* Patients with ischemic stroke within one week;
* Patients with Bronchial asthma, Chronic obstructive pulmonary disease (COPD), and patients with diseases related to dyspnoea;
* Any contraindication against the use of ticagrelor and other study drugs;
* Platelet count less than 100 x 109/L;
* Haemoglobin (Hb) level less than 100 g/L;
* Researchers involved in the study and / or immediate family members;
* Participation in another investigation drug or device study in the past 30 days before enrollment;
* Involvement in the planning and conduct of the study (applies to staffs at study sites);
* Suffering from other serious disorders and the life expectancy less than half year;
* Increased risk of bradycardic events (e.g. no pacemaker and known sick sinus syndrome, second degree A-V block, third degree A-V block or previous documented syncope suspected to be due to bradycardia). The Sponsor will review the Holter data in this study to assess the need to continue with this exclusion;
* Pregnancy or lactation or females of child-bearing potential with the plan of pregnancy in one year;
* Concomitant oral or intravenous therapy (see examples below) with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers which cannot be stopped for the course of the study （Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir; Substrates with narrow therapeutic index: cyclosporine, quinidine；Strong inducers: rifampin/rifampicin, phenytoin, carbamazepine).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Overall bleeding events | 18 months

SECONDARY OUTCOMES:
Major bleeding events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Genshan Ma, PhD., Study Director — Southeast University; Yu Wang, MD., Principal Investigator — Southeast University; Yuyu Yao, Ph.D, Principal Investigator — Southeast University; Wenbin Lu, MD., Principal Investigator — Southeast University; Cong Fu, MD., Principal Investigator — Southeast University; LIjuan Chen, PhD., Principal Investigator — Southeast University
Locations (3):
- China (3):
  - Zhongda Hospital, Nanjing, Jiangsu
  - The forth hospital of Xuzhou, Xuzhou, Jiangsu
  - Jiangbin hospital, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu W, Wang Y, Chen L, Li Y, Zhang R, Chen Z, Yan J, Yang M, Han B, Wang Z, He S, Chen L, Wu X, Zeng H, Ma L, Shi G, Yin J, Chen J, Ma G. Antithrombotic Therapy With Ticagrelor in Atrial Fibrillation Subjects After Percutaneous Coronary Intervention. Front Cardiovasc Med. 2021 Oct 12;8:745549. doi: 10.3389/fcvm.2021.745549. eCollection 2021. PMID 34712714
- [Derived] Lu W, Chen L, Wang Y, Yao Y, Fu C, Zuo P, Ma G. Rationale and design of MANJUSRI trial: a randomized, open-label, active-controlled multicenter study to evaluate the safety of combined therapy with ticagrelor and warfarin in AF subjects after PCI-eS. Contemp Clin Trials. 2015 Jan;40:166-71. doi: 10.1016/j.cct.2014.12.002. Epub 2014 Dec 13. PMID 25513965